CLINICAL TRIAL: NCT01998919
Title: A Randomised, Placebo-controlled, Double-blind Phase II of Sequential Administration of Tarceva (Erlotinib) or Placebo in Combination With Gemcitabine/Platinum as First-line Treatment in Patients With Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC).
Brief Title: A Study of Tarceva (Erlotinib) in Combination With Platinum Based Chemotherapy in Patients With Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MO18633
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tarceva + gemcitabine/platinum (Experimental)
  Interventions: Drug: erlotinib [Tarceva]; Drug: gemcitabine; Drug: cisplatin; Drug: carboplatin
- Placebo + gemcitabine/platinum (Placebo Comparator)
  Interventions: Drug: placebo; Drug: gemcitabine; Drug: cisplatin; Drug: carboplatin

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg orally daily Days 15 to 28 of each 4-week cycle for 6 cycles, followed by 150 mg orally daily
  Arms: Tarceva + gemcitabine/platinum
Drug: placebo — orally daily Days 15 to 28 of each 4-week cycle for 6 cycles, followed by daily oral application
  Arms: Placebo + gemcitabine/platinum
Drug: gemcitabine — 1250 mg/m2 iv Days 1 and 8 of each 4-week cycle, 6 cycles
Drug: cisplatin — 75 mg/m2 iv Day 1 of each 4.wek cycle, 6 cycles; or carboplatin
Drug: carboplatin — 5 x AUC iv Day 1 of each 4.week cycle, 6 cycles; or cisplatin

SUMMARY:
This study will evaluate the efficacy and safety of sequential administration of Tarceva and gemcitabine/platinum chemotherapy in patients with stage IIIb/IV non-small cell lung cancer. Patients will be randomized to receive Tarceva (150 mg po) or placebo on days 15-28 of a 4 week cycle of intravenous platinum-based chemotherapy, for a total of 6 cycles. The anticipated time on study treatment is until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically documented advanced or recurrent stage IIIB or IV non-small cell lung cancer;
* measurable disease;
* no previous chemotherapy for non-small cell lung cancer.

Exclusion Criteria:

* unstable systemic disease;
* any other malignancies in the last 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2006-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (14):
- Australia (3):
  - Campbelltown
  - Camperdown
  - Liverpool
- China (2):
  - Guangzhou
  - Shanghai
- Hong Kong, Hong Kong
- Indonesia (3):
  - Jakarta
  - Semarang
  - Yogyakarta
- Philippines (2):
  - Manila
  - Metro Manila
- Kyunggi-do, South Korea
- Taipei, Taiwan
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Plus Chemotherapy: Participants received placebo tablets, orally (PO), on Days 15 to 28 of a 4-week cycle; participants also received platinum-based doublet chemotherapy: gemcitabine 1250 milligrams per square meter (mg/m^2) via intravenous (IV) infusion on Days 1 and 8 and either cisplatin (75 mg/m^2) or carboplatin (5 times [x] area under the serum concentration-time curve [AUC]), via IV infusion, per investigator discretion, on Day 1. Participants received study drugs for a maximum of 6 cycles until disease progression, unacceptable toxicity or death. After 6 cycles, participants may have continued to receive placebo tablets daily.
- Erlotinib Plus Chemotherapy: Participants received erlotinib tablets, 150 mg per day, PO on Days 15 to 28 of every 4-week cycle; participants also received platinum-based doublet chemotherapy: gemcitabine 1250 mg/m^2 via IV infusion on Days 1 and 8 and either cisplatin (75 mg/m^2) or carboplatin (5 x AUC), via IV infusion, per investigator discretion, on Day 1. Participants received study drugs for a maximum of 6 cycles until disease progression, unacceptable toxicity or death. After 6 cycles, participants may have continued to receive erlotinib monotherapy, 150 mg daily.
Period: Overall Study
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Started | 79 | 74
Randomized | 78 (1 participant randomized to erlotinib didn't receive study drug; analyzed in placebo for safety) | 76 (One participant withdrew consent prior to 1st dose and was excluded from safety analysis population.)
Completed | 37 | 39
Not Completed | 42 | 35
Not completed — Death | 2 | 2
Not completed — Adverse Event | 0 | 5
Not completed — Disease progression | 31 | 22
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all randomized participants. For analysis, participants were assigned the treatment group to which they were randomized, regardless of the treatment they actually received.
Groups:
- Placebo Plus Chemotherapy: Participants received placebo tablets, PO, on Days 15 to 28 of a 4-week cycle; participants also received platinum-based doublet chemotherapy: gemcitabine 1250 mg/m^2 via intravenous (IV) infusion on Days 1 and 8 and either cisplatin (75 mg/m^2) or carboplatin (5 x AUC), via IV infusion, per investigator discretion, on Day 1. Participants received study drugs for a maximum of 6 cycles until disease progression, unacceptable toxicity or death. After 6 cycles, participants may have continued to receive placebo tablets daily.
- Total: Total of all reporting groups
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy | Total
Number analyzed (Participants) | 78 | 76 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.06) | 56.4 (10.43) | 56.45 (10.245)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non-Progression at Week 8 as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Non-progression defined as documented best overall tumor response of complete response (CR), partial response (PR), or stable disease (SD; where SD was maintained for greater than [>]8 weeks) per RECIST. Investigator's assessment of response used in all analyses. CR equals (=)disappearance of all target lesions; PR=at least a 30 percent (%) decrease in sum of longest diameter (LD) of target lesions, taking as reference the baseline sum LD; SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference smallest sum LD since treatment started.
Time Frame: Week 8
Population: FAS; for analysis, participants were assigned the treatment group to which they were randomized, regardless of the treatment they actually received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo Plus Chemotherapy: Participants received placebo tablets, PO, on Days 15 to 28 of a 4-week cycle; participants also received platinum-based doublet chemotherapy: gemcitabine 1250 mg/m^2 via IV infusion on Days 1 and 8 and either cisplatin (75 mg/m^2) or carboplatin (5 x AUC), via IV infusion, per investigator discretion, on Day 1. Participants received study drugs for a maximum of 6 cycles until disease progression, unacceptable toxicity or death. After 6 cycles, participants may have continued to receive placebo tablets daily.
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 78 | 76
percentage of participants | 76.9 [66.0 to 85.7] | 80.3 [69.5 to 88.5]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; Mean Difference (Final Values) = 3.34, 95% CI 2-sided [-10.3 to 17.0] — Approximate 95% CI for difference of two rates using Hauck-Anderson method

2. Secondary Outcome: Percentage of Participants With Non-Progression at Week 16 as Assessed by RECIST
Description: Non-progression defined as documented best overall tumor response of CR, PR, or SD (where SD was maintained for >16 weeks) per RECIST.
Time Frame: Week 16
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 78 | 76
percentage of participants | 53.8 [42.2 to 65.2] | 64.5 [52.7 to 75.1]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; Mean Difference (Final Values) = 10.63, 95% CI 2-sided [-5.6 to 26.8] — Approximate 95% CI for difference of two rates using Hauck-Anderson method

3. Secondary Outcome: Percentage of Participants With Confirmed CR or PR as Assessed by RECIST
Description: CR=disappearance of all target lesions; PR=at least a 30% decrease in sum of LD of target lesions, taking as reference the baseline sum LD.
Time Frame: Screening/Baseline, Day 22 of Cycles 2, 4 and 6 and every 8 weeks in Post-Study and Off-Study Phases
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 78 | 76
percentage of participants | 24.4 [15.3 to 35.4] | 36.8 [26.1 to 48.7]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; Mean Difference (Final Values) = 12.48, 95% CI 2-sided [-2.7 to 27.7] — Approximate 95% CI for difference of two rates using Hauck-Anderson method

4. Secondary Outcome: Duration of Response
Description: Duration of Response was defined similarly for complete responders and partial responders. CR was defined as the date CR was first recorded to the date on which PD was first noted or date of death. PR was defined as the date the first PR was recorded to the date of the first observation of PD or date of death.
Time Frame: Screening/Baseline, Day 22 of Cycles 2, 4 and 6 and every 8 weeks in Post-Study and Off-study Phases
Population: FAS; only participants with CR or PR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 19 | 28
weeks | 24.1 [17 to 33] | 38.4 [25 to 77]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.0075, Log Rank
Statistical Analysis 2: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.0099, Wald test; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.22 to 0.81]

5. Secondary Outcome: Time to Progression
Description: Time to progression was defined as the interval between the day of randomization and the first documentation of PD. Participants who were withdrawn from the study without documented progression and for whom there exists CRF evidence that evaluations have been made, were censored at 1) the date of the last tumor assessment, 2) last date in the drug log, or 3) last date of follow-up when the participant was known to be progression free, whichever was last. Participants without post-baseline tumor assessments but known to be alive were censored at the time of randomization.
Time Frame: Screening/Baseline, Day 22 of Cycles 2, 4 and 6 and every 8 weeks in Post-Study and Off-Study Phases
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 78 | 76
weeks | 24.1 [18 to 28] | 31.4 [25 to 36]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.0004, Log Rank
Statistical Analysis 2: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.0001, Wald Test; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.33 to 0.70]

6. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the interval between the day of randomization and the date of first documentation of progressive disease or date of death, whichever came first.
Time Frame: Screening/Baseline, Day 22 of Cycles 2, 4 and 6 and every 8 weeks in Post-Study and Off-Study Phases
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 78 | 76
weeks | 23.4 [17 to 25] | 30.4 [24 to 34]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.0001, Log Rank
Statistical Analysis 2: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p < 0.0001, Wald test; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.33 to 0.68]

7. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment.
Time Frame: Date of randomization until date of death or date of last follow-up assessment
Population: FAS Population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Number analyzed (Participants) | 78 | 76
weeks | 75.7 [60 to 105] | 74.1 [49 to 100]
Statistical Analysis 1: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.5991, Log Rank
Statistical Analysis 2: Comparison: Placebo Plus Chemotherapy vs Erlotinib Plus Chemotherapy; Test type: Superiority or Other; p = 0.3774, Wald test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.58 to 1.23]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout primary and post-study treatment phases and for 28 days after last study dose.
Description: The Safety Analysis Population (SAP) included all participants who received at least 1 dose/infusion and had at least 1 post-baseline safety assessment. For analysis, participants were assigned to the treatment group of the first received dose irrespective of subsequent changes in treatment.
Arm/Group | Placebo Plus Chemotherapy | Erlotinib Plus Chemotherapy
Serious Adverse Events (participants affected / at risk) | 17/79 | 17/74
Other Adverse Events (participants affected / at risk) | 74/79 | 73/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Chemotherapy (N=79) | Erlotinib Plus Chemotherapy (N=74)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Plus Chemotherapy (N=79) | Erlotinib Plus Chemotherapy (N=74)
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 10
Nausea (Gastrointestinal disorders) | 37 | 34
Vomiting (Gastrointestinal disorders) | 29 | 22
Constipation (Gastrointestinal disorders) | 25 | 22
Diarrhoea (Gastrointestinal disorders) | 20 | 26
Stomatitis (Gastrointestinal disorders) | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 3 | 5
Mouth ulceration (Gastrointestinal disorders) | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 33 | 30
Fatigue (General disorders) | 18 | 23
Pyrexia (General disorders) | 11 | 10
Chest pain (General disorders) | 10 | 5
Asthenia (General disorders) | 5 | 5
Mucosal inflammation (General disorders) | 1 | 6
Anaemia (Blood and lymphatic system disorders) | 12 | 19
Neutropenia (Blood and lymphatic system disorders) | 17 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6
Leukopenia (Blood and lymphatic system disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 11 | 9
Platelet count decreased (Investigations) | 5 | 7
White blood cell count decreased (Investigations) | 7 | 5
Neutrophil count decreased (Investigations) | 5 | 6
Haemoglobin decreased (Investigations) | 4 | 6
Dizziness (Nervous system disorders) | 6 | 7
Dysgeusia (Nervous system disorders) | 2 | 5
Neuropathy peripheral (Nervous system disorders) | 1 | 4
Paronychia (Infections and infestations) | 0 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Renal impairment (Renal and urinary disorders) | 4 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 4
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Dry mouth (Gastrointestinal disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 32 | 48
Acne (Skin and subcutaneous tissue disorders) | 2 | 8
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 9
Malaise (General disorders) | 7 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Alanine aminotransferase increased (Investigations) | 8 | 3
White blood cell count (Investigations) | 6 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 2
Neutrophil count (Investigations) | 4 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Headache (Nervous system disorders) | 9 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2
Hypertension (Vascular disorders) | 4 | 3
Tinnitus (Ear and labyrinth disorders) | 4 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic lesion (Hepatobiliary disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Wound (Injury, poisoning and procedural complications) | 0 | 1
Breast swelling (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 3
Vision blurred (Eye disorders) | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 2
Abnormal sensation in eye (Eye disorders) | 1 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1
Eye pain (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Vein pain (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 1 | 1
Nail infection (Infections and infestations) | 0 | 2
Oral herpes (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tinea infection (Infections and infestations) | 0 | 1
Tinea versicolour (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 3 | 1
Somnolence (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Blood creatinine increased (Investigations) | 2 | 1
Platelet count (Investigations) | 2 | 1
Blood sodium decreased (Investigations) | 1 | 1
Haemoglobin (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 2 | 0
Weight decreased (Investigations) | 1 | 1
Weight increased (Investigations) | 1 | 1
Alanine aminotransferase (Investigations) | 1 | 0
Aspartate aminotransferase (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Blood creatinine abnormal (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Neutrophil percentage decreased (Investigations) | 0 | 1
Sputum abnormal (Investigations) | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 3
Pain (General disorders) | 3 | 2
Chills (General disorders) | 2 | 2
Influenza like illness (General disorders) | 2 | 2
Oedema peripheral (General disorders) | 1 | 2
Oedema (General disorders) | 2 | 0
Catheter site swelling (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Local swelling (General disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Gastritis (Gastrointestinal disorders) | 0 | 3
Glossitis (Gastrointestinal disorders) | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.